CLINICAL TRIAL: NCT04414085
Title: The Clinical Significance of Biochemical Polymorphism in the 11 Deoxycortisol Levels Before and After Stimulation With Adrenocorticotrofin
Brief Title: The Clinical Significance of Biochemical 11 Deoxycortisol Levels
Status: Completed | Type: Observational
Sponsor: Assaf Harofeh MC (Other Government)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Galia Askapa, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 0183-15-ASF
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Retrospective

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
data from charts regarding clinical characteristics and androgens levels from first to last visit were collected

DETAILED DESCRIPTION:
data from charts regarding clinical characteristics and androgens levels from first to last visit were collected Female patients only ages 10-18 years who were referred to the combined gynecology endocrinology adolescents clinic

ELIGIBILITY:
Inclusion Criteria:

age 10-18 years referred to gynecology endocrinology adolescents clinic

Exclusion Criteria:

no data available in chart no blood work available

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: All referred to gynecology endocrinology adolescents clinic who underwent an ACTH stimulation test
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Presence of hyperandrogenism signs (1 to 3 categorized) | 3 years
  hirsuitism, acne, menses, each marked as 0 or 1 (none or present)

CONTACTS AND LOCATIONS:
Overall Officials: galia barash, md, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Undecided